CLINICAL TRIAL: NCT04749602
Title: A Phase II Trial of Intrapleural Instillation of the Nivolumab in Cancer Patients With Pleural Effusion.
Brief Title: Intrapleural Instillation of the Nivolumab in Cancer Patients With Pleural Effusion.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCRB-Hadassah-01
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Renal Cell Cancer Metastatic; Non-small Cell Lung Cancer Metastatic; Pleural Effusion, Malignant
Keywords: Nivolumab; Intrapleural irrigation; Pleural carcinomatosis
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Cohort 1 (renal cell carcinoma / lung cancer) Cohort 2 (lung cancer)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Intrapleural Nivolumab in patients with renal cell carcinoma (Experimental): Drainage followed by nivolumab (40 mg, single intrapleural instillation) will be performed.
  Interventions: Drug: Nivolumab
- Cohort 2: Intrapleural Nivolumab in patients with non-small cell lung cancer (Experimental): Drainage followed by nivolumab (40 mg, single intrapleural instillation) will be performed.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — 40 mg of the nivolumab will be used intrapleurally (once).
  Other Names: Opdivo

SUMMARY:
Patients with advanced cancers who have pleural effusion, especially those requiring pleural evacuation, experienced poorer survival when treated with immunotherapy. The pleura also acts as a natural barrier that can limit the penetration of immune checkpoint inhibitors. In this multicenter phase 2 study, the preliminary efficacy and toxicity of intrapleural instillation of the nivolumab in patients with immune-sensitive metastatic cancers will be accessed.

DETAILED DESCRIPTION:
Patients ≥18 years old who have large volume of pleural effusion, required evacuation, and received systemic therapy with a checkpoint inhibitor (monotherapy or combination with another checkpoint inhibitor) for metastatic cancers (renal cell carcinoma (RCC) and non-small cell lung cancer (NSCLC) will be eligible. Drainage followed by nivolumab (40 mg, single intrapleural instillation) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Large volume of pleural effusion (1 liter and more), required evacuation
* Systemic therapy with a checkpoint inhibitor (monotherapy or combination with another checkpoint inhibitor)
* Metastatic cancers (renal cell carcinoma (RCC) and non-small cell lung cancer (NSCLC)

Exclusion Criteria:

* Autoimmune disorders
* Previous treatment for

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
3-month recurrence-free survival | 3 months
  Proportion of patients who will be without signs of radiographic recurrence after 3 months

SECONDARY OUTCOMES:
Rate of any grade adverse events | 3 months
  Percentage of patients who will experience any grade adverse events (according to CTCAE criteria ver. 5.0) associated with intrapleural nivolumab use

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Tsimafeyeu, M.D., Principal Investigator — Kidney Cancer Research Bureau
Locations (5):
- Russia (5):
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - Kidney Cancer Research Bureau, Moscow
  - Medicine 24/7 clinic, Moscow
  - Medscan, Moscow
  - Yauza clinical hospital, Moscow